CLINICAL TRIAL: NCT06533436
Title: Clinical and Economic Comparison of 2 Methods of Intubation Tube Fixation in the Intensive Care Unit: Benefits of Intubation Tube Fixation with AnchorFastTM Versus Current Cord Fixation
Brief Title: Clinical and Economic Comparison of 2 Methods of Intubation Tube Fixation : AnchorFastTM Versus Current Cord Fixation
Acronym: AnchorDon
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2021_0208; 2023-A01371-44 (Other: ANSM)
Record Dates: First submitted 2024-02-28; First posted 2024-08-01 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Intubation Complication; Eschar

STUDY DESIGN:
Intervention Model Description: A total of 170 patients will be included over two distinct 6-month periods (85 patients per period). Each period corresponds to the study of one fixation device: cord fixation or fixation with the AnchorFastTM medical device.
  The caregivers will also be included as a population since the workload with the two types of device will be evaluated and compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cord attachement (Active Comparator): Caregivers follow the Tensoplast® white cord and elastic plaster fixation protocol, which has been revised and validated by the care department.
  Tube care is carried out in two stages: preparing the patient for the procedure (safety and hygiene) then renewal of the fixation device.
  Interventions: Procedure: Corded tube care
- AnchorFast (Experimental): The AnchorFastTM fixation device developed by Laboratoire Hollister is a single-use medical device. This fixation system consists of a hard plastic guide on which the intubation tube can slide laterally.
  It facilitate access to the oral cavity and limit pressure points on the corners of the mouth.
  Interventions: Device: Tube care attached by AnchorFast
- Caregivers (Other): The caregivers will be included as a study population. Caregivers will conduct the search for the other two arms (ancofast and by cord) and then fill in questionnaires assessing the workload and comfort of tube care.
  Interventions: Other: Caregiver's evaluation on each tube fixation

INTERVENTIONS:
Procedure: Corded tube care — The caregiver cut a 6 cm strip of Tensoplast® and wrapped it around the intubation probe at the level of the prescribed fixation mark at the corner of the mouth. The cord strands are placed around the patient's head, tightened, and a double knot is tied at the patient's cheek. Compresses are placed over the ears to protect them from possible lesions caused by the cords.
  Arms: Cord attachement
Device: Tube care attached by AnchorFast — Shaving is recommended for patients with beards, and prior family consent is required for patients with beards.
  AnchorFast is Suitable for intubation probes from 5 to 10 mm in diameter, it adapts to different morphologies thanks to hydrocolloid dressings bonded to the face and an adjustable cord around the neck. Due to its rigidity, this device is not recommended for patients whose condition requires them to be positioned in the ventral decubitus (VD) or lateral decubitus position.
  Arms: AnchorFast
Other: Caregiver's evaluation on each tube fixation — The caregivers who performs the interventions according to the study will fill question form to assess the worload and the confort of the tube care for each intervention type The caregivers are both a research actor and a study population. One of the secondary aims of this study is to evaluate the two types of tube-fixing with regard to caregiver workload and comfort in performing care. Caregivers will complete identical questionnaires assessing their satisfaction with the two types of tube fixation studied in arms 1 and 2.
  Arms: Caregivers

SUMMARY:
The aim of this study is to assess the benefits of using the Anchorfast device in reducing complications associated with intubation tube fixation, in terms of the rate of pressure ulcer development, the rate of intubation tube mobilization and the rate of VAP occurrence. If the hypothesis is confirmed, this project would enable the caregivers to optimize the current practice in the interests of both patients and caregivers. That's why the investigators have designed a real-life study, and will also be looking at the effect of care load on and caregiver satisfaction.

DETAILED DESCRIPTION:
In 2022 at Hôpital FOCH, 41% of patients admitted to the intensive care unit required an orotracheal intubation tube (OIT), exposing them to the risk of developing orotracheal intubation tube (OIT), exposing them to the risk of developing ventilator-associated pneumonia (VAP).

Preventing VAP involves oral hygiene and limiting tube movements, which depend on the device used to attach the OIT . The care protocol used routinely in the department uses adhesive tape and a rigid cotton haberdashery cord. This type of fixation impedes buccal access, prevents easy repositioning of the probe and is liable to cause eschar lesions.

With the aim of improving the practices, the investigators took a closer look at the French recommendations. The Société de Réanimation de Langue Française (French Intensive Care Society) does not recommend a particular fixation method, but it does relay publications that shows the superiority of the AnchorfastTM device over adhesive tape fixation in terms of the incidence of pressure sores and accidental catheter mobilization.

The aim of this study is to assess the benefits of using the Anchorfast device in reducing complications associated with intubation tube fixation, in terms of the rate of pressure ulcer development, the rate of intubation tube mobilization and the rate of VAP occurrence. If the hypothesis is confirmed, this project would enable the caregivers to optimize the current practice in the interests of both patients and caregivers. That's why the investigators have designed a real-life study, and will also be looking at the effect of care load on and caregiver satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old,
* Patient with orotracheal intubation,
* Patient intubated no more than 24 hours previously,
* Oral consent from patient, trusted support person or relative if unable to consent
* Membership of a French health insurance scheme.

Exclusion Criteria:

* Pre-existing facial, labial or auricular skin lesions,
* Pre-existing mucositis,
* Patients extubated for more than 24 hours whose condition requires a new intubation tube
* Nasotracheal intubation,
* Planned early tracheotomy,
* Patient with occipital craniectomy,
* Patient in ventral position,
* Pregnant or breast-feeding woman,
* Patient deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2026-08-02 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of induced pressure sores | 16 months
  Evaluate the change in the incidence rate of eschars (grade 1 or higher according to the National Pressure Ulcer Advisory Panel 1998 classification) induced by fixation of the intubation tube with the AnchorFastTM device compared with the cord fixation cord fixation technique.

SECONDARY OUTCOMES:
Patient safety regarding the stability of the intubation : number of repositionning | 16 months
  Compare tube attachment stability between the 2 groups : Every day, as part of routine care for intubated patients, the correct position of the tube is recorded and checked. Each repositioning of the intubation tube is also recorded.
Patient safety regarding the risk of accidental extubation | 16 months
  Compare the number of accidental extubation between the 2 groups
Patient safety regarding ventilator-associated pneumonia | 16 months
  Compare the rate of ventilator-associated pneumonia (VAP) between the 2 groups
Patient safety regarding intubation-related complications | 16 months
  Evaluate the occurrence of intubation-related complications
Impact on nursing staff care load | 16 months
  Comparing the care load between the 2 groups (Nursing Activity Score) . The scale comprises 7 categories for a total of 23 items: basic activities (monitoring and controls, laboratory tests, medication, hygiene measures, drain care, mobilization and positioning, support and accompaniment of families and patients, administrative and management tasks), respiratory assistance, cardiovascular assistance, renal assistance, neurological assistance, metabolic assistance and specific interventions.
  The final score is expressed as a percentage of nursing time.
Impact on nursing staff comfort according to the Nursing Activity Score. | 16 months
  Compare the comfort of use of the device by nursing staff during the provision of care between the 2 groups The scale comprises 7 categories for a total of 23 items: basic activities (monitoring and controls, laboratory tests, medication, hygiene measures, drain care, mobilization and positioning, support and accompaniment of families and patients, administrative and management tasks), respiratory assistance, cardiovascular assistance, renal assistance, neurological assistance, metabolic assistance and specific interventions.
  The final score is expressed as a percentage of nursing time.
Budgetary impact : comparison of the average total price per patient (consumables, labor), taking into account additional expenses in the event of medical complications related to the fixation system | 16 months
  Carry out a comparative budget impact analysis : The costs of each method of intubation tube fixation will be calculated per patient, in order to perform a medico-economic analysis. The following will be measured: the cost of consumables in each group, the cost of adverse events (PAVM, accidental extubation, etc.) and the cost of nursing time allocated to this management.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa LAGOA PINTO, Principal Investigator — Hôpital Foch
Locations (1):
- Hôpital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No